CLINICAL TRIAL: NCT06680479
Title: Safety and Immunogenicity of Stabilized CH505 TF chTrimer Vaccination in Adults Living With HIV-1 on Suppressive Antiretroviral Therapy
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Temporarily Closed (paused)
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Duke University (Other); Access to Advanced Health Institute (AAHI) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5422; 39037 (Other: DAIDS-ES ID)
Record Dates: First submitted 2024-11-07; First posted 2024-11-08 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: HIV-1
Keywords: HIV; Therapeutic vaccine; bNab-inducing vaccine; Trimer
MeSH Terms: interventions — Sodium Chloride; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Randomized (2:1), 20 participants in Arm 1 and 10 participants in Arm 2
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Study Arm 1: CH505 TF chTrimer (300 mcg) admixed with 3M-052-AF (3 mcg) and Alum (500 mcg) (Experimental)
  Interventions: Biological: CH505 TF chTrimer; Biological: 3M-052-AF; Biological: Aluminum Hydroxide Suspension
- Study Arm 2: Placebo (sodium chloride for injection, 0.9% USP) (Placebo Comparator)
  Interventions: Other: Sodium Chloride for Injection

INTERVENTIONS:
Biological: CH505 TF chTrimer — Stabilized CH505 TF chTrimer, 300 mcg
  Arms: Study Arm 1: CH505 TF chTrimer (300 mcg) admixed with 3M-052-AF (3 mcg) and Alum (500 mcg)
Biological: 3M-052-AF — 3 mcg
  Arms: Study Arm 1: CH505 TF chTrimer (300 mcg) admixed with 3M-052-AF (3 mcg) and Alum (500 mcg)
Biological: Aluminum Hydroxide Suspension — 500 mcg
  Arms: Study Arm 1: CH505 TF chTrimer (300 mcg) admixed with 3M-052-AF (3 mcg) and Alum (500 mcg)
Other: Sodium Chloride for Injection — Sodium chloride for injection, 0.9% USP volume-matched placebo injection.
  Arms: Study Arm 2: Placebo (sodium chloride for injection, 0.9% USP)

SUMMARY:
A5422 is a phase 1, randomized, double-blind, placebo-controlled clinical trial to assess the safety, tolerability, and immunogenicity of a vaccination with stabilized CH505 TF chTrimer admixed with 3M-052-AF + Aluminum hydroxide (Alum), to assess the effect of CH505 TF chTrimer vaccine as a therapeutic vaccine in adults living with HIV-1 on suppressive antiretroviral therapy (ART) with the aim of inducing new HIV-1 Envelope (Env) B-cell neutralizing immune responses. Participants will be on study for up to 100 weeks (52 weeks on study treatment plus 48 weeks follow-up).

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* On a suppressive ART regimen for at least 24 months with no changes in the 90 days prior to study entry
* CD4+ cell count greater than 200 cells/mm3 obtained within 56 days prior to study entry
* HIV-1 RNA <200 copies/mL obtained within 56 days prior to study entry
* Plasma HIV-1 RNA levels <200 copies/mL for at least 12 months on ART prior to study entry
* The following laboratory values obtained within 56 days prior to study entry

  * White blood cell count ≥2,500 cells/mm3
  * Absolute neutrophil count (ANC) >750/mm3
  * Hemoglobin ≥11 g/dL for cisgender men/transgender women and ≥10 g/dL for cisgender women/transgender men
  * Platelet count ≥100,000/mm3
  * Creatinine <1.5x upper limit of normal (ULN)
  * Alanine aminotransferase (ALT) (SGPT) ≤1.5 ULN
* Hepatitis C Virus (HCV) antibody-negative or HCV RNA negative result if indicated, within 56 days prior to study entry
* Negative hepatitis B surface antigen (HBsAg) result obtained within 56 days prior to study entry
* For study candidates of child-bearing potential, negative serum or urine pregnancy test at screening and within 48 hours prior to study entry
* No participation in conception process and agree to use at least one reliable form of contraception if participating in sexual activity that could lead to pregnancy during the study and for 8 weeks following the final study vaccine

Exclusion Criteria:

* Known to have started ART during acute HIV infection
* Known to have HIV-related opportunistic infections within the last 2 years prior to study entry.
* History of malignancy within the last 5 years prior to study entry.
* Currently breastfeeding
* History of or active autoimmune disorders
* HIV vaccination (prophylactic and/or therapeutic) within 1 year prior to study entry
* Receipt of any anti-HIV-1 bNAbs within 2 years prior to study entry
* Vaccination within 4 weeks prior to study entry
* Use of any infusion blood product or immune globulin within 16 weeks prior to study entry (Exception: COVID-19-specific monoclonal antibodies are allowed)
* Use of systemic immunomodulators, systemic cytotoxic chemotherapy, or non-FDA approved investigational therapy within 60 days prior to study entry
* Intent to use immunomodulators during the course of the study
* Immune deficiency other than HIV
* HCV antiviral therapy within 90 days prior to screening
* Known allergy/sensitivity or any hypersensitivity to components of study drug(s) or their formulation
* Active drug or alcohol use or dependence that would interfere with adherence to study requirements
* Acute or serious illness requiring systemic treatment and/or hospitalization within 30 days prior to study entry
* Conditions that would preclude injection site reaction assessments (e.g., extensive tattoos, scarring, skin conditions).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-04-14 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who initiated active study treatment (CH505 TF chTrimer, 3M-052-AF and Alum) who met the study-defined primary safety composite endpoint | Day 0 (after initial vaccination) to 4 weeks (28 days) after the last vaccination
  The study-defined primary safety endpoint is a composite endpoint. A participant who has initiated active study treatment is considered to have met the endpoint if the participant has experienced any treatment-related (i.e., related to CH505 TF chTrimer, 3M-052-AF or Alum as judged by the core team, blinded to study treatment) 1) serious adverse event (SAE), or 2) Grade 3+ adverse event (AE), or 3) AE that led to permanent discontinuation of study treatment regardless of grade
Number of the viruses with antibody neutralization response for a cross-clade global panel of 9 viruses expressing heterologous envelopes determined using a neutralization assay | Day 0 pre-vaccination to 2 weeks (14 days) after the fifth vaccination

SECONDARY OUTCOMES:
Antibody neutralization response for vaccine-matched and related viruses | Day 0 pre-vaccination to 2 weeks (14 days) after the fifth vaccination
  Determined using a neutralization assay and CH505 TF and related vaccine matched virus panel

CONTACTS AND LOCATIONS:
Overall Officials: Madhu Choudhary, MD, Study Chair — University of Pittsburgh
Locations (25):
- United States (25):
  - University of California, Los Angeles CARE Center CRS, Los Angeles, California
  - UCSD Antiviral Research Center CRS, San Diego, California
  - University of California, San Francisco HIV/AIDS CRS, San Francisco, California
  - Harbor University of California Los Angeles Center CRS, Torrance, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - The Ponce de Leon Center CRS, Atlanta, Georgia
  - Northwestern University CRS, Chicago, Illinois
  - Johns Hopkins University CRS, Baltimore, Maryland
  - Massachusetts General Hospital CRS (MGH CRS), Boston, Massachusetts
  - Washington University Therapeutics (WT) CRS, St Louis, Missouri
  - New Jersey Medical School Clinical Research Center CRS, Newark, New Jersey
  - Weill Cornell Chelsea CRS, New York, New York
  - Columbia Physicians & Surgeons (P&S) CRS, New York, New York
  - Weill Cornell Uptown CRS, New York, New York
  - University of Rochester Adult HIV Therapeutic Strategies Network CRS, Rochester, New York
  - Chapel Hill CRS, Chapel Hill, North Carolina
  - Greensboro CRS, Greensboro, North Carolina
  - Cincinnati CRS, Cincinnati, Ohio
  - Case CRS, Cleveland, Ohio
  - Ohio State University CRS, Columbus, Ohio
  - Penn Therapeutics CRS, Philadelphia, Pennsylvania
  - University of Pittsburgh CRS, Pittsburgh, Pennsylvania
  - Vanderbilt Therapeutics (VT) CRS, Nashville, Tennessee
  - Houston Advancing Research Team CRS, Houston, Texas
  - University of Washington Positive Research CRS, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the AIDS Clinical Trials Group by NIH.
Access Criteria: * With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the AIDS Clinical Trials Group.
  * For what types of analyses? To achieve aims in the proposal approved by the AIDS Clinical Trials Group.
  * By what mechanism will data be made available? Researchers may submit a request for access to data using the AIDS Clinical Trials Group "Data Request" form at: https://actgnetwork.org/submit-a-proposal/. Researchers of approved proposals will need to sign an AIDS Clinical Trials Group Data Use Agreement before receiving the data.